CLINICAL TRIAL: NCT05835596
Title: MumCare: Mum's Cardiovascular Health for Life
Acronym: MumCare
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian SIDS and Stillbirth Society (Other); University of Oslo (Other)
Responsible Party: Principal Investigator, Anne Cathrine Staff, Professor and Head of research (Div. Obst and Gyn), Oslo University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 478376
Record Dates: First submitted 2023-03-08; First posted 2023-04-28 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Hypertensive Disorder of Pregnancy; Preeclampsia; Gestational Hypertension; Gestational Diabetes
MeSH Terms: conditions — Toxemia; Pre-Eclampsia; Hypertension, Pregnancy-Induced; Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: Women are ranomized to MumCare app access or not for the 14-18 month intervention time
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Access to MumCare app (Active Comparator): Women will be randomized prospectively (before or after delivery) after they consent to participate in the study. These women are at increased risk of longterm cardiovascular disease due to hypertensive or gestational diabetes pregnancy complication. This group is randomized to have access to the MumCare app will, in addition to standard care, have access to the app for 14-18 months following giving birth. The MumCare app has 3 main parts (1. an educational part, 2. The patient's own health data (entered by the user herself) that represent modifiable risk factors for cardiovascular disease), and 3. The app will send push reminders for the woman to book a visit at her general practitioner according to recommended guidelines (that are usually not followed-up today).
  All women in the study will be invited to a cardiovascular health evaluation at 14-18 months postpartum.
  Interventions: Device: Access to MumCare app
- No access to MumCare app (No Intervention): Women will be prosepctively randomized (before or after delivery) after they consent to participate in the study. These women are at increased risk of longterm cardiovascular disease due to hypertensive or gestational diabetes pregnancy complication. Women randomized to NOT have access to the MumCare app will receive standard care, which includes being provided oral and written information according to delivery ward routines.
  All women in the study will be invited to a cardiovascular health evaluation at 14-18 months postpartum.

INTERVENTIONS:
Device: Access to MumCare app — Education, push warning to book cardiovascular health follow-up at own general practitioner , registration of BP and lipids, HbAc
  Arms: Access to MumCare app

SUMMARY:
The goal of this randomized clinical trial study is to test the potential benefits of eHealth-assisted follow-up after pregnancy complications that confer and increased risk for premature cardiovascular (CV) disease.

The overarching aim is to improve short- and long-term CV health in women following pregnancy complications associated with increased risk of CV disease (hypertensive disorders of pregnancy and gestational diabetes). The investigators will develop and test a novel, personalized and user co-designed digital eHealth companion ("app") and test the app in a clinical randomized control trial. The group randomized to app use will get access to the app prior to delivery or within the first weeks postpartum, whereas the control group will not get access to the app, but receive ordinary follow-up. Both groups are invited to a comprehensive cardiovascular follow-up 14-18 months post delivery.

The primary objective is to assess whether the rate of 1-year postpartum follow-up at the general practitioner's is increased with MumCare app access. Secondary objectives are to assess:

1. expectations of (and satisfaction with) postpartum eHealth-assisted technologies,
2. if health perception, sense of empowerment, quality of life, modifiable risk factors for CV disease (including hypertension, dyslipidemia, blood sugar control, smoking, weight), CV findings (including non-invasive hemodynamics) and biomarkers are affected by MumCare app use.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is a leading cause of premature death and morbidity in women. CVD prevention is most effective when started at subclinical stages. Preeclampsia, gestational hypertension, and gestational diabetes are female sex-specific risk factors for CVD. Postpartum follow-up programs for the primary prevention of CVD following these complications are not offered today. In the MumCare study, a randomized control trial (RCT) will test a new eHealth app that promotes a personalized cardiovascular (CV) health optimization in young women after such pregnancy complications.

The study will first assess users' expectations of eHealth-assisted follow-up following the aforementioned pregnancy complications. These users will test and help fine-tune the new MumCare app, which integrates patient self-registered health data with an educational follow-up program based on Norwegian obstetric - and the Norwegian Directorate of Health guidelines. The study will recruit women to use the MumCare app in a 1:1 RCT lasting 18 months postpartum. App use (in the active study arm) will be registered in secure IT systems.

The primary outcome for comparison between groups (women with and without app access) is the rate of 1-year postpartum follow-up with a general practitioner (as recommended in the obstetric guidelines). Secondary outcomes include user-reported outcomes (such as health empowerment and quality of life) and objective risk factors for CVD (evaluated 14-18 months postpartum in all study groups, including assessment of CV risk factors, CV function and biomarkers).

ELIGIBILITY:
Inclusion Criteria:

* An ongoing or recent pregnancy complicated by hypertensive disorder of pregnancy and/or gestational diabetes mellitus
* Patient attending Oslo University Hospital, Oslo, Norway
* Signed informed written consent (to be randomized to app access or not)

Exclusion Criteria:

* Not capable of accessing and using an app downloaded on a smart phone
* Not able to understand the informed consent or app instructions or content (in Norwegian, but later the study consent form and app will be translated into English and other languages)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
General Practitioner attendance 1 year postpartum | 1 year postpartum
  Cardiovascular risk screening at general practitioner attendance (guideline recommeded, but rarely followed-up by patients)

SECONDARY OUTCOMES:
Patient Reported Outcome Measures (PROM); SF-36 | 13-14 months postpartum
  Patient reported (by online questionnaires) health-related quality of life (short-form-health survey 36).
  The Short-Form Health Survey 36 (SF36) scale consists of 36 items related to health perception, grouped into eight multi-item scales ranging from 0 to 100 (0=worst, 100=best). Differences in SF-36 subscale scores of 5 points have been considered clinically relevant.
Patient Reported Outcome Measures (PROM); heiQ | 13-14 months postpartum
  Patient reported (by online questionnaires) health-related quality of life: health education impact questionnaire.
  The Health Education Impact Questionnaire (heiQ) scale consists of 40 items representing 8 domains that evaluates immediate effects of self-management interventions. Items are scored on a scale ranging from 1 (strongly disagree) to 4 (strongly agree), higher score in the heiQ scales indicates better status, except for "emotional distress", where higher score indicates higher distress.
Patient Reported Outcome Measures (PROM); GSE | 13-14 months postpartum
  Patient reported (by online questionnaires) health-related quality of life: general self-efficacy scale.
  The General Self Efficacy (GSE) Scale measures optimistic self-beliefs in coping with the challenges of life. : "refers to optimistic self-beliefs of being able to perform and control behaviors, and is linked with various physical and mental health outcomes". Responses on 10 items are reported on a four point scale ranging from 1 (not at all true) to 4 (exactly true). The score of the total scale ranges from 10 to 40, higher score indicates higher GSE.
Patient Reported Outcome Measures (PROM); SOC-13 | 13-14 months postpartum
  Patient reported (by online questionnaires) health-related quality of life: sense of coherence.
  The Sense of Coherence (SOC-13) scale consists of 13 items measuring the perception of manageability, meaningfulness and comprehensibility. The scale of the items ranges from 1 to 7, while the total sum ranges from 13 to 91, where higher score indicates a higher sense of coherence.
Patient Reported Outcome Measures (PROM); EPDS | 13-14 months postpartum
  Patient reported (by online questionnaires) health-related quality of life: Edinburgh Postnatal Depression Scale.
  The Edinburgh Postnatal Depression Scale (EPDS) scale consists of 10 items evaluating depression on a total score from 0 to 30. A score of ≥10 indicates depression.
Qualitative interviews of users and their General Practiotioner | 13-14 montths postpartum
  Compare user experiences (health perception, empowerment, quality of life) with and without app use (for both woman and her GP)
Clinical cardiovascular follow-up at recruitment hospital: Blood pressure | 14-18 months postpartum
  Normotension (or not) at 14-18 months postpartum (blood pressure below 140 mmHg systolic AND below 90 mmHg diastolic)
Clinical cardiovascular follow-up at recruitment hospital: BMI | 14-18 months postpartum
  Normal weight (or not) at 14-18 months postpartum; defined as body mass index (weight in kilo s divided by height in square meters) below 25 kg/m2
Clinical cardiovascular follow-up at recruitment hospital: HbA1c | 14-18 months postpartum
  Normal HbA1(or not) at 14-18 months postpartum; defined as below 42 mmol/L. Diabetes mellitus is diagnosed if HbA1c is 48 mmol/L or above, whereas HbA1c of 42-47 mmol/L indicates high risk for developing diabetes (and life style intervention combined with annual HbA1c assessment is therefore recommended)
Clinical cardiovascular follow-up at recruitment hospital: HDL | 14-18 months postpartum
  Normal (or not) level of high density lipoprotein at 14-18 months postpartum; defined as HDL of 1.3 mmol/L or above (for women). HDL below 1.3 mmol/L indicates high risk for developing cardiovascular disease.
Clinical cardiovascular follow-up at recruitment hospital: Total cholesterol | 14-18 months postpartum
  Normal (or not) level of total serum cholesterol at 14-18 months postpartum; defined as serum cholesterol at or below 5 mmol/L. Total cholesterol above 5 mmol/L indicates increased risk for developing cardiovascular disease. Total cholesterol of or above 7 mmol/L indicates most often therapy.
Clinical cardiovascular follow-up at recruitment hospital: LDL cholesterol | 14-18 months postpartum
  Normal (or not) level of LDL (low density lipoprotein) cholesterol at 14-18 months postpartum; defined as LDL cholesterol at or below 3 mmol/L. LDL cholesterol above 3 mmol/L indicates increased risk for developing cardiovascular disease. LDL cholesterol of or above 5 mmol/L indicates most often therapy.
Clinical cardiovascular follow-up at recruitment hospital: fTG | 14-18 months postpartum
  Normal (or not) level of fasting serum triglycerides at 14-18 months postpartum; defined as fTG at or below 1.7 mmol/L. fTG above 1.7 mmol/L combined with HDL cholesterol below 1.2 mmol/L in women indicates dyslipidemia and increased risk for developing cardiovascular disease.
Clinical cardiovascular follow-up at recruitment hospital: ApoB | 14-18 months postpartum
  Normal (or not) serum Apolipoptotein B at 14-18 months postpartum; defined as ApoB above 1.4 g/L. The normal reference range for women is 0.5-1.4 g/L.
  High levels indicate increased risk for developing cardiovascular disease.
Clinical cardiovascular follow-up at recruitment hospital: Apo A1 | 14-18 months postpartum
  Normal (or not) serum Apolipoptotein A1 at 14-18 months postpartum; defined as Apo A1 within the normal reference range for women: 1.1-2.0 g/L.
Clinical cardiovascular follow-up at recruitment hospital: ApoB/Apo A1 ratio | 14-18 months postpartum
  Normal (or not) serum Apolipoptotein B/Apolipoprotein A1 ratio at 14-18 months postpartum; defined as ApoB/Apo A1 ratio at or below 0.6.
  In women, a ratio above 0.6 indicates increased risk of cardiovascular disease.
Clinical cardiovascular follow-up at recruitment hospital: waist-hip-ratio | 14-18 months postpartum
  Normal (or not) waist to hip ratio (both measured in same unit; in nearest full cm) at 14-18 months postpartum; defined as a ratio below 0.85 in women.
Clinical cardiovascular follow-up at recruitment hospital: waist circumference | 14-18 months postpartum
  Normal (or not) waist circumference (measured in nearest full cm) at 14-18 months postpartum; defined as a below 88 cm in women.
Clinical cardiovascular follow-up at recruitment hospital: serum biomarkers associated to cardiovascular risk | 14-18 months postpartum
  Compare serum cardiovascular biomarker levels (between the 2 study groups) at a general cardiovascular health assessment at 14-18 months postpartum. Following (elevated levels) biomarkers have been associated with increased cardiovascular risk, and will be assessed for group comparison following study finalization:
  hsCRP, high-sensitive C-reactive protein GDF-15, growth differentiation factor 15 sHLA-G, soluble human leukocyte antigen G cTnT, cardiac-specific high sensitive Troponin T NT-proBNP, n-terminal pro-brain natriuretic peptide SAA1, serum amyloid 1

CONTACTS AND LOCATIONS:
Overall Officials: Anne Cathrine Staff, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
Only data that alone or in combination cannot identify a unque patient will be shared, that is at group level, in accordance with patient consent and IRB approval in Norway.